CLINICAL TRIAL: NCT04082286
Title: 90Yttrium-labelled Anti-CD66 Monoclonal Antibody as Part of a Reduced Intensity Conditioning Regimen Prior to Allogeneic Haematopoietic Stem Cell Transplantation: an Open Label, Dose Escalating Phase I Study in Children and Adolescents With Relapsed/Refractory Leukaemia
Brief Title: Yttrium-90 Anti CD66 Monoclonal Antibody in Childhood Relapsed/Refractory Leukaemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07MI05
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2020-10

CONDITIONS: Acute Myeloblastic Leukemia; Acute Lymphoblastic Leukemia; Juvenile Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Juvenile | interventions — Radioimmunotherapy

STUDY DESIGN:
Intervention Model Description: 3+3 Dose escalation study, patient will receive 111In-labelled anti-CD66 MoAb (dosimetry) and 90Yttrium-labelled anti-CD66 MoAb (for therapy)
Masking Description: Yttrium-90 labelled monoclonal antibody against CD66
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radioimmunotherapy (Experimental): Children affected by high risk malignant disorders will be receiving increasing infused activity of a radio-immune conjugated antibody as part of their conditioning regimen prior to alleogeneic stem cell transplantation
  Interventions: Other: Yttrium-90 labelled monoclonal antibody against CD66

INTERVENTIONS:
Other: Yttrium-90 labelled monoclonal antibody against CD66
  Other Names: Radioimmunotherapy

SUMMARY:
The radio-labeled anti-CD66 monoclonal antibody (with 111In for dosimetry and 90Y for therapy) will be administered in the T11 North room, UCLH, while the reduced intensity conditioning regimen and the allogeneic hematopoietic stem cell transplant will be performed in 2 centers, according to the age of the patient: A) patients aged < 13 years will be transplanted at the Bone Marrow Transplantation Department, Great Ormond Street Hospital (GOSH), and B) patients aged 13-18 years will be transplanted at the Bone Marrow Transplantation Department, University College London Hospitals (UCLH).

ELIGIBILITY:
Inclusion criteria:

1. An underlying haematological malignancy including:

   1. isolated bone marrow relapse of AML after allogeneic haematopoietic stem cell transplantation;
   2. isolated bone marrow relapse of ALL after allogeneic haematopoietic stem cell transplantation;
   3. bone marrow relapse of JMML after allogeneic haematopoietic stem cell transplantation;
   4. refractory AML (5-20% blasts in BM) with/without expression of CD66 on blasts;
   5. refractory ALL (5-20% blasts in BM) with/without expression of CD66 on blasts;
   6. refractory AML (> 20% blasts in BM) with expression of CD66 on blasts;
   7. refractory ALL (> 20% blasts in BM) with expression of CD66 on blasts;
2. be ≥ 1 year old and ≤ 18 years old;
3. must not be eligible for therapy of higher curative potential. Where an alternative therapy has been shown to prolong survival in an analogous population, this should be offered to the patient prior to discussing this study;
4. have a Karnofsky Performance Status ≥ 50 or Lansky Performance Status ≥ 30;
5. provide signed, written informed consent from parent or guardian;
6. be able to comply with study procedures and follow-up examinations;
7. have normal cardiac function without specific treatment;
8. have adequate organ function (as indicated by Table 3, chapter 5), within 30 days prior to 111In infusion;
9. patients who have received any other chemotherapy within the previous 2 weeks and must have recovered from acute toxicity of all previous therapy prior to enrolment;
10. be negative for human-anti-murine antibodies (HAMA). Exclusion criteria

1) patients with CNS disease; 2) patients with BM cellularity < 10%; 3) patients with ≥ 20% blasts in BM and no expression of CD66 on blasts; 4) patients who are positive for human-anti-murine antibodies (HAMA); 5) patients with compromised organ function (as indicated by Table 3, chapter 5), within 30 days prior to 111In infusion; 6) patients with extensive chronic GvHD; 7) patients with an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment; 8) patients who are pregnant or lactating; 9) patients with any other severe concurrent disease, which, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 45 days post transplant
  targeted radiotherapy delivered by 90Yttrium-labelled anti-CD66
dose limited toxicity (DLT) | 45 days post transplant
  targeted radiotherapy delivered by 90Yttrium-labelled anti-CD66

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital for Children, London, United Kingdom